CLINICAL TRIAL: NCT07335900
Title: A Clinical Study Using FAPI-PET Imaging to Evaluate the Effects of TAVI on Reversing Myocardial Structural and Functional Remodeling in Patients With Aortic Stenosis
Brief Title: A Clinical Study Using FAPI-PET Imaging to Assess the Postoperative Effects of TAVI in Patients With Aortic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IIT-2025-0364
Record Dates: First submitted 2025-12-26; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Severe Aortic Valve Stenosis
Keywords: Severe aortic valve stenosis; Transcatheter Aortic Valve Replacement; FAPI-PET
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVI+OMT (Experimental): Patients in the TAVI group will undergo transcatheter aortic valve implantation according to standard clinical procedures and receive optimal medical therapy.
  Interventions: Procedure: Transcatheter Aortic Valve Implantation; Drug: Optimal medication treatment
- OMT (Other): Optimal medication treatment
  Interventions: Drug: Optimal medication treatment

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Implantation — Patients in the TAVI group underwent transcatheter aortic valve implantation performed by the hospital's cardiac intervention team according to standard clinical procedures, and received optimal medical therapy（The recommended medications include: First category: SGLT2 inhibitors (gliflozin drugs) such as dapagliflozin and empagliflozin; Second category: Angiotensin receptor-neprilysin inhibitors (ARNI) with the representative drug sacubitril/valsartan; Third category: β-blockers (the '-lol' class) with representative drugs including bisoprolol, metoprolol sustained-release tablets, and carvedilol; Fourth category: Mineralocorticoid receptor antagonists (MRA, aldosterone receptor antagonists) with representative drugs spironolactone and eplerenone; Fifth category (for specific populations): vericiguat. Diuretics should be individualized, including loop diuretics such as furosemide and torasemide.）.
  Arms: TAVI+OMT
Drug: Optimal medication treatment — All enrolled patients must receive the Optimal medication treatment（The recommended medications include: First category: SGLT2 inhibitors (gliflozin drugs) such as dapagliflozin and empagliflozin; Second category: Angiotensin receptor-neprilysin inhibitors (ARNI) with the representative drug sacubitril/valsartan; Third category: β-blockers (the '-lol' class) with representative drugs including bisoprolol, metoprolol sustained-release tablets, and carvedilol; Fourth category: Mineralocorticoid receptor antagonists (MRA, aldosterone receptor antagonists) with representative drugs spironolactone and eplerenone; Fifth category (for specific populations): vericiguat. Diuretics should be individualized, including loop diuretics such as furosemide and torasemide.）.

SUMMARY:
This study will include patients with severe degenerative aortic stenosis (AS) who meet the inclusion criteria and voluntarily participate (planned to undergo TAVI), as well as patients with aortic stenosis who have not undergone valve replacement (control group). All enrolled patients will undergo a ^18F-FAPI-1801 PET/CT scan at baseline (before or at the time of TAVI) and 6 months postoperatively to quantitatively evaluate myocardial fibroblast activation and structural remodeling indicators, and to follow up on changes in clinical cardiac function. Patients with aortic stenosis receiving only medical therapy will be set as the control group for comparative analysis, to assess the impact of relieving aortic stenosis on the reduction of myocardial fibrosis activity, myocardial remodeling, and reversal of cardiac function.

ELIGIBILITY:
Inclusion Criteria:

① Age 18 years or older, any gender; ② Confirmed diagnosis of severe degenerative aortic stenosis by echocardiography (valve area AVA < 1.0 cm² or mean transvalvular gradient > 40 mmHg; for AS with reduced ejection fraction and low-flow, low-gradient, the presence of outflow tract reserve must be confirmed with dobutamine stress); ③ Evaluated by the heart team as unsuitable for surgical open-heart valve replacement due to advanced age or severe comorbidities, without anatomical contraindications, and expected to benefit from transcatheter valve implantation. Patients who meet these criteria and decide to undergo TAVI will be assigned to the TAVI group; those who meet the criteria but do not undergo valve replacement will enter the control group (possible scenarios include: relatively mild valve stenosis not meeting TAVI indication, or patient refusal of surgery, opting for drug therapy only, etc.).

Exclusion Criteria:

* Recent acute myocardial infarction (less than 1 month from onset to enrollment) or the presence of active myocarditis, infectious endocarditis, and other acute inflammatory conditions, as these conditions can significantly affect FAPI uptake and cardiac function; ② History of old myocardial infarction (with existing myocardial scarring and remodeling, which affect fibroblast imaging); ③ Presence of uncontrolled severe arrhythmias, such as persistent ventricular tachycardia, ventricular fibrillation, or high-risk second-degree or higher atrioventricular block, resulting in hemodynamic instability due to arrhythmia within the past 3 months; ④ Concomitant severe cardiovascular diseases affecting study evaluation, including severe valvular disease (excluding AS, such as severe mitral regurgitation), hypertrophic obstructive cardiomyopathy, primary pulmonary hypertension, etc.; ⑤ Presence of examination contraindications: allergy to PET tracers or MRI contrast agents, severe renal insufficiency (eGFR <30 ml/min/1.73 m²) with inability to tolerate gadolinium-enhanced MRI, or severe claustrophobia preventing compliance with imaging examinations; ⑥ Allergic constitution (history of allergy to multiple drugs or unknown substances); ⑦ Pregnant or breastfeeding women (female subjects of childbearing potential must provide a negative pregnancy test before enrollment and use effective contraception during the study); ⑧ Any other situation that the investigator believes could significantly increase study risk or interfere with result interpretation, such as active malignant tumors or advanced disease with expected survival of less than 1 year; ⑨ Inability to comply with the trial protocol or follow-up requirements (e.g., poor prior adherence, expected inability to attend scheduled follow-ups).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
FAPI-PET myocardial uptake value | Baseline and 6 months after enrollment
  All enrolled patients underwent a ^18F-FAPI-1801 PET/CT scan at baseline (before or at the time of TAVI) and at 6 months postoperatively to quantitatively assess the degree of myocardial fibroblast activation and structural remodeling indicators, with follow-up on clinical cardiac function changes. Patients with aortic stenosis who received only medical treatment were set as a control group for comparative analysis to evaluate the effect of relieving aortic stenosis on reducing myocardial fibrosis activity, as well as on myocardial remodeling and reversal of cardiac function.

CONTACTS AND LOCATIONS:
Overall Officials: Jun PU, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital,Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided